CLINICAL TRIAL: NCT02907580
Title: Influenza Vaccine Attitudes, Intent, and Receipt
Brief Title: Influenza Vaccine Attitudes, Intent, and Receipt: Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, Associate Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAQ9636
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Vaccination; Influenza
Keywords: influenza; vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Local educational data (Experimental): Local-based educational handout
  Interventions: Behavioral: Local educational information
- National educational data (Experimental): National-based educational handout
  Interventions: Behavioral: National educational information
- Usual care (No Intervention): No educational information other than provided as usual care by health care providers

INTERVENTIONS:
Behavioral: Local educational information — Participants in this arm receive educational information regarding influenza vaccination based on local educational information.
  Arms: Local educational data
Behavioral: National educational information — Participants in this arm receive educational information regarding influenza vaccination based on national educational information.
  Arms: National educational data

SUMMARY:
Influenza vaccine is recommended as routine care for all individuals who are at least 6 months of age and older. Recently, questions about vaccine safety and concerns for side effects have increased, contributing to both influenza vaccine hesitancy and refusal. In an effort to educate parents and patients, public health entities and physicians give informational handouts in various forms. However, recent publications have found that pro-vaccine messages can have paradoxical effects on vaccine intentions, therefore further studies on vaccine related public health communication is needed. Few, if any, studies have analyzed the relationship between influenza vaccine attitudes and intention with actual vaccine receipt in the pediatric population. These results will help to understand the relationship between parent's vaccine perception and the intent to vaccinate versus the child's receipt of the influenza vaccine, as well as to optimize educational information given to families regarding the influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 6 months

Exclusion Criteria:

* Receipt of influenza vaccination that season

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Number of children who receive influenza vaccination on day of intervention | Day 0
  Receipt of influenza vaccination by the child on the day of the educational intervention

SECONDARY OUTCOMES:
Number of children who receive influenza vaccination during the influenza vaccine season | Up to 7 months
  Receipt of influenza vaccination by the child by April 2017
Number of parents who anticipate influenza vaccination during the influenza vaccine season | Up to 7 months
  Parents report planned receipt of influenza vaccination by themselves by April 2017

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scott VP, Opel DJ, Reifler J, Rikin S, Pethe K, Barrett A, Stockwell MS. Office-Based Educational Handout for Influenza Vaccination: A Randomized Controlled Trial. Pediatrics. 2019 Aug;144(2):e20182580. doi: 10.1542/peds.2018-2580. Epub 2019 Jul 10. PMID 31292219